CLINICAL TRIAL: NCT04736147
Title: A Phase 1 Open-label Study to Assess the Immunogenicity, Safety, and Reactogenicity of JNJ-64300535, a DNA Vaccine Administered by Electroporation-mediated Intramuscular Injection, in Healthy Participants
Brief Title: A Study of JNJ-64300535 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108950; 2020-005277-27 (EudraCT Number); 64300535HPB1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JNJ-64300535 (Experimental): Participants will receive an electroporation-mediated intramuscular (IM) injection of JNJ-64300535 vaccine.
  Interventions: Biological: JNJ-64300535

INTERVENTIONS:
Biological: JNJ-64300535 — JNJ-64300535 injection will be administered intramuscularly.

SUMMARY:
The purpose of this study is to evaluate the cellular immunogenicity of 3 monthly electroporation-mediated intramuscular (IM) injections of JNJ-64300535 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) indicating that he understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Must be healthy as confirmed by medical history, physical examination, and vital signs performed at screening

Exclusion Criteria:

* Weight of less than (<) 50 kilograms (kg) and a body mass index (BMI) <19.0 or greater than (>) 29.9 kilogram per meter square (kg/m^2) at screening
* History of Human Immunodeficiency Virus (HIV) infection or a positive HIV antibody test at screening
* History of HBV infection, measured by the presence of HBsAg and/or anti-HBc antibodies
* History of seizure disorders unless seizure free for >5 years
* Has a non-removable active electronic stimulation device

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Responding Against Hepatitis B Virus (HBV) Core or Polymerase (Pol) Vaccine Antigens | Up to Day 67
  Percentage of participants responding against HBV Core or Pol vaccine antigens will be reported.

SECONDARY OUTCOMES:
Number of Participants With Solicited Local Adverse Events (AEs) | Up to Day 64
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs are pre-defined local (at the injection site) AEs for which participants will be specifically questioned and which will be noted by participants in their diary for 7 days post first vaccination. Solicited local AEs are: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site.
Number of Participants With Solicited Systematic Adverse Events | Up to Day 64
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants will be instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events will include fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Number of Participants With Serious Adverse Events (SAEs) | Up to Day 225
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with SAEs will be reported.
Number of Participants With Unsolicited Adverse Events | Up to Day 225
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are events which will be reported by the participant voluntarily or obtained by means of interviewing the participant in a non-directed manner at study visits.
Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Up to Day 225
  Number of participants with clinically significant abnormalities in laboratory parameters such as (hematology, blood biochemistry, blood coagulation and urinalysis) will be reported.
Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) | Up to Day 113
  Number of participants with clinically significant abnormalities in ECG will be reported.
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Up to Day 225
  Number of participants with clinically significant abnormalities in vital signs (including body temperature, pulse/heart rate, systolic and diastolic blood pressure) will be reported.
Number of Participants With Clinically Significant Abnormalities in Physical Examination | Up to Day 225
  Number of participants with clinically significant abnormalities in physical examination (including height, body weight, skin examination, and other body systems) will be reported.
Percentage of Participants With a Positive T-cell Response Against HBV Core or Pol Vaccine Antigens | Up to Day 225
  Percentage of participants with a positive T-cell response against HBV Core or Pol vaccine antigens will be reported.
Breadth of the T-cell Responses Against HBV Core or Pol Vaccine Antigens | Up to Day 225
  Breadth of the T-cell responses against HBV Core or Pol vaccine antigens will be reported.
Magnitude of the T-cell Responses Against HBV Core or Pol Vaccine Antigens | Up to Day 225
  Magnitude of the T-cell responses against HBV Core or Pol vaccine antigens will be reported
Number of Cytokines of Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) T-cell Responses Against HBV Core or Pol Vaccine Antigens | Up to Day 225
  Number of cytokines of both CD4 and CD8 T-cell responses against HBV Core or Pol vaccine antigens will be reported.
Frequency of Intramuscular TriGrid Delivery System version 2.0 (TDS-IM v2.0) Device Faulty Conditions | Up to Day 57
  Frequency of device fault conditions observed during administration of study treatment with TDS-IM v2.0 device will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Verheijden S, Conceicao-Neto N, Bourgeois S, Vandamme C, Troyer E, Kanoulas E, Maeyer D, Crabbe M, Makariadou E, Slaets L, Fevery B, Remoortere PV, Biermer M, Kennedy PTF, De Creus A. Safety, immunogenicity, and baseline immune correlates of vaccine JNJ-0535 in participants with or without CHB. NPJ Vaccines. 2026 Feb 5. doi: 10.1038/s41541-025-01364-x. Online ahead of print. PMID 41644953